CLINICAL TRIAL: NCT04437875
Title: An Open Study of the Safety, Tolerability and Immunogenicity of the Drug "Gam-COVID-Vac Lyo" Lyophilizate for the Preparation of a Solution for Intramuscular Injection With the Participation of Healthy Volunteers
Brief Title: An Open Study of the Safety, Tolerability and Immunogenicity of "Gam-COVID-Vac Lyo" Vaccine Against COVID-19
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Collaborators: Acellena Contract Drug Research and Development (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 03-Gam-COVID-Vac Lyo-2020
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-06

CONDITIONS: Preventive Immunization COVID-19
Keywords: COVID-19; SARS-CoV-2; vector vaccine; adenovirus vector
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: An open, prospective, two-stage, non-randomized, first-phase study involving healthy volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Component 1 (Experimental): rAd26 Component, 1 vaccination Component 1 consists of a recombinant adenovirus vector based on the human adenovirus type 26, containing the SARS-CoV-2 S protein gene.
  Interventions: Biological: Gam-COVID-Vac Lyo
- Component 2 (Experimental): rAd5 Component, 1 vaccination Component 2 consists of a vector based on the human adenovirus type 5, containing the SARS-CoV-2 S protein gene.
  Interventions: Biological: Gam-COVID-Vac Lyo
- Prime-Boost Immunization (Experimental): Day 1 rAd26 Component Day 21 rAd5 Component
  Interventions: Biological: Gam-COVID-Vac Lyo

INTERVENTIONS:
Biological: Gam-COVID-Vac Lyo — adenoviral-based vaccine against SARS-CoV-2

SUMMARY:
the purpose of this study: to evaluate the safety, tolerability and immunogenicity of the drug "Gam-COVID-Vac Lyo", a lyofilizate for preparing solution for intramuscular administration, at various times after vaccination in healthy adult volunteers.

DETAILED DESCRIPTION:
An open two stage non-randomized Phase 1 study with the participation of healthy volunteers. This clinical trial is an open study of safety, tolerability and immunogenicity of the drug "Gam-COVID-Vac Lyo", lyophilisate for the preparation of a solution for intramuscular administration, with the participation of healthy volunteers.

Study objectives

1. A safety and tolerability assessment of the drug "Gam-COVID-Vac Lyo", lyophilisate for the preparation of a solution for intramuscular administration, using single dose of each component (Stage 1).
2. A safety and tolerability assessment of the drug "Gam-COVID-Vac Lyo", lyophilisate for the preparation of a solution for intramuscular administration, using prime-boost immunization according to the proposed scheme (Stage 2).

Study Design Stage 1 the First group, 9 volunteers, will receive the drug, a solution for intramuscular administration, in the mode of single immunization with component 1 in a full therapeutic dose.

the Second group, 9 volunteers, will receive the drug, a solution for intramuscular administration, in the mode of single immunization with component 2 in the full therapeutic dose.

The studied drugs will be administered to a total of 18 volunteers in a hospital setting and after administration, the drug's safety will be continuously monitored for 5 days. Based on the results of the safety assessment, the Chief investigator decides to proceed to the second stage of the study on the 5th day after the introduction of the studied drugs.

Second stage The second stage will include 20 volunteers and three understudies. Volunteers of the second stage will be vaccinated no earlier than 5 days after vaccination of participants of the first stage.

Volunteers participating in the second stage of the study (a total of 20 people) will receive the study drug according to the booster scheme: the introduction of component 1 will be carried out on day 1, and component 2-on the 21st day of the study. Follow-up will be carried out during 4 visits: on 7, 14, 28, 42 days after administration of the drug.

Throughout the inpatient observation and the follow-up period (180 days) of visits during the entire study, safety information will be collected

ELIGIBILITY:
Inclusion Criteria:

1. males and females within the age range from 18 to 60 years;
2. written informed consent;
3. subject body mass index (BMI): 18.5 ≤ BMI ≤ 30;
4. negative PCR test results for SARS-CoV-2 (during the screening);
5. no history of COVID-2019 disease;
6. no contacts of volunteers with patients with COVID-2019 for at least 14 days;
7. negative test results for IgM and IgG antibodies to SARS-CoV-2;
8. subject agrees to use effective contraceptive methods during the entire period of participation in the study;
9. absence of acute infectious diseases at the time of vaccine administration and 14 days before vaccination;
10. negative pregnancy test of blood or urine (for women of childbearing age);
11. subject has negative tests for HIV, hepatitis B and С, syphilis or confirmed medical history;
12. subject has a negative result of the urine test for residual narcotic drugs;
13. negative test for alcohol in exhaled air;
14. the absence of malignant diseases of any nature and localization;
15. in medical history and based on the screening results, subject has no diseases or pathologies of the gastrointestinal system, liver, kidneys, cardiovascular system and blood, CNS, musculoskeletal system, urogenital, immune and endocrine systems that from the point of view of the researcher and/or of the organizer of the study, may affect the safety of the volunteer and the evaluation of the study results (clinical, instrumental and laboratory tests did not reveal diseases or clinically significant deviations)

Exclusion Criteria:

1. volunteer involvement in another study over the last 90 days;
2. any vaccination over the last 30 days;
3. history of COVID-2019 disease;
4. positive PCR test results for SARS-CoV-2 (during the screening);
5. positive test results for IgM and IgG antibodies to SARS-CoV-2;
6. health staff in contact with people with COVID-2019;
7. respiratory symptoms in the last 14 days;
8. the administration of immunoglobulins or other blood products in the last 3 months;
9. regular current or past use of narcotic drugs;
10. subject has received immunosuppressive and/or immunomodulating agents within 6 months before the start of the study;
11. pregnancy or breast feeding;
12. exacerbation of allergic diseases at the time of vaccination;
13. subject has systolic blood pressure less than 100 mm Hg or greater than 139 mm Hg; diastolic blood pressure less than 60 mm Hg or greater than 90 mm Hg; heart rate lower than 60 beats per minute or above 100 beats per minute;
14. a burdened allergic history (anaphylactic shock, Quincke's edema, polymorphic exudative eczema, atopy, a history of serum sickness, hypersensitivity or allergic reactions to the introduction of any vaccines in history, known allergic reactions to vaccine components, etc.);
15. a history of autoimmune diseases in the volunteer's medical history and in relatives' medical history of the 1-2 degree of kinship;
16. subject smokes more than 10 cigarettes per day;
17. alcohol intake exceeding the low-risk level: no more than 20 grams of pure alcohol per day, no more than 5 days a week, alcohol intake within 48 hours before the administration of the drug;
18. planned hospitalization and/or surgery during the period of participation in the study, as well as 4 weeks before the expected date of the administration of the drug;
19. the presence of an associated disease that may affect the assessment of the results of the study;
20. any conditions that, according to the researcher's doctor, may be a contraindication to the participation in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
The changing of antibody levels against the SARS-CoV-2 glycoprotein S at 42 days | at days 0, 14, 21, 28, 42
  Determination of antibody levels against the SARS-CoV-2 glycoprotein S measured by an ELISA vs. baseline values
Number of Participants With Adverse Events | through the whole study, an average of 180 days
  Determination of Number of Participants With Adverse Events

SECONDARY OUTCOMES:
The changing of virus neutralizing antibody titer | at days 0, 14, 28, 42
  Determination of virus neutralizing antibody titer
The changing of antigen-specific cellular immunity level | at days 0, 14, 28
  Determination of antigen-specific cellular immunity (specific T-cell immunity, in particular, IFN-gamma production or lymphoproliferation)

CONTACTS AND LOCATIONS:
Overall Officials: Lola Morozova, Md, Principal Investigator — I.M. Sechenov First Moscow State Medical University
Locations (1):
- Sechenov First Moscow State Medical University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Logunov DY, Dolzhikova IV, Zubkova OV, Tukhvatullin AI, Shcheblyakov DV, Dzharullaeva AS, Grousova DM, Erokhova AS, Kovyrshina AV, Botikov AG, Izhaeva FM, Popova O, Ozharovskaya TA, Esmagambetov IB, Favorskaya IA, Zrelkin DI, Voronina DV, Shcherbinin DN, Semikhin AS, Simakova YV, Tokarskaya EA, Lubenets NL, Egorova DA, Shmarov MM, Nikitenko NA, Morozova LF, Smolyarchuk EA, Kryukov EV, Babira VF, Borisevich SV, Naroditsky BS, Gintsburg AL. Safety and immunogenicity of an rAd26 and rAd5 vector-based heterologous prime-boost COVID-19 vaccine in two formulations: two open, non-randomised phase 1/2 studies from Russia. Lancet. 2020 Sep 26;396(10255):887-897. doi: 10.1016/S0140-6736(20)31866-3. Epub 2020 Sep 4. PMID 32896291